CLINICAL TRIAL: NCT01396902
Title: Text Reminders for Immunization Compliance in Kids
Brief Title: Text Reminders for Immunization Compliance in Kids (TRICKS) Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Carolyn R. Ahlers-Schmidt, PhD, Associate Research Professor, University of Kansas
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-018
Record Dates: First submitted 2011-07-17; First posted 2011-07-19 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Child Immunizations
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator)
  Interventions: Behavioral: Standard of care
- Text Messaging (Experimental)
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Standard of care — You will receive an immunization handout and verbal instructions regarding your child's next apt. Your child's immuniztion records will also be checked through KSWebIZ an internet based system that tracks immunizations for kids in Kansas.
  Arms: Standard of care
Behavioral: Text Messaging — You will receive text message reminders prior to your child's two, four and six month immunization due dates. You will be asked to take part in a phone interview and your child's immuniztion records will be checked through KSWebIZ an internet based system that tracks immunizations for kids in Kansas.
  Arms: Text Messaging

SUMMARY:
As a participant in these research program you will be a parent of a child born at Wesley Medical Center who plan to use Carriage Park Pediatric Clinic for your child's care. Mobile phone text messages will be sent to remind you of your child's immunizations.

The long term research goal is to increase childhood immunization rates by improving parental health literacy through an innovative text messaging system regarding immunization schedules for children under the age of six.

ELIGIBILITY:
Inclusion Criteria:

* parent or caregiver of a well child born at Wesley Medical Center;
* planning to utilize the Carriage Park Pediatric Clinic for his/her child's medical home; (
* adult (> 18 years of age);
* present use of a mobile phone for sending and receiving text messages;
* English or Spanish speaking;
* able to provide informed consent.

Exclusion criteria include:

* personal or religious beliefs against immunizations;
* inability to complete enrollment information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
the first aim is to assess our ability to enroll at least 70% (N=90) of eligible parents in a text messaging program | up to 1 year
  This will be accomplished through recruitment of parents of newborns at Wesley Medical Center who will receive care from Carriage Park Clinic.

SECONDARY OUTCOMES:
the second aim is to implement the TRICKs intervention with parents of newborns. | up to 1 year
  SMSCaster software will be assessed for its ability to send appointment reminders and to collect follow-up data from parents regarding whether immunization appointments were scheduled.
the third aim is to collect immunization information on participant's children. | up to 1 year
  This will be accomplished using the Kansas Immunization Registry (KSWebIZ), a web-based centralized birth to death database that maintains complete, accurate, and secure immunization records for all Kansas residents.

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas University School of Medicine-Wichita, Wichita, Kansas, United States

REFERENCES:
- [Derived] Ahlers-Schmidt CR, Chesser AK, Nguyen T, Brannon J, Hart TA, Williams KS, Wittler RR. Feasibility of a randomized controlled trial to evaluate Text Reminders for Immunization Compliance in Kids (TRICKs). Vaccine. 2012 Aug 3;30(36):5305-9. doi: 10.1016/j.vaccine.2012.06.058. Epub 2012 Jun 29. PMID 22750044